CLINICAL TRIAL: NCT06004791
Title: A Prospective, Randomized, Controlled Study of rhTPO in Combination With Herombopag + CsA vs Herombopag + CsA for the Treatment of Primary Transfusion-dependent NSAA
Brief Title: A Prospective, Randomized, Controlled Study of rhTPO in Combination With Herombopag + CsA vs Herombopag + CsA for the Treatment of Primary TD-NSAA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rHCsA
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Aplastic Anemia; Drug Effect
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herombopag + CsA (Placebo Comparator): Herombopag 10mg/ day, adjust the dose according to the blood image, the course of treatment is at least 3 months, CsA: 3-5 mg/kg/d, adjust the valley concentration 100-200ng/ml, at least 6 months, effective patients continue to use for 1 year, and then gradually reduce the dose.
  Interventions: Drug: Herombopag + CsA
- rhTPO combined with Herombopag + CsA (Experimental): Administer rhTPO (15000U, subcutaneously once daily for 7 days, once a month for 3 months),Herombopag 10mg/day, adjust dose according to blood picture for at least 3 months, CsA: 3-5 mg/kg/d, adjust trough concentration 100-200ng/ml for at least 6 months, continue for 1 year if effective, then gradually reduce dose
  Interventions: Drug: rhTPO combined with Herombopag + CsA

INTERVENTIONS:
Drug: Herombopag + CsA — Herombopag（10mg/d）+CsA(3-5 mg/kg/d, adjust the grain concentration 100-200ng/ml)
  Other Names: control
  Arms: Herombopag + CsA
Drug: rhTPO combined with Herombopag + CsA — rhTPO (15000U, subcutaneous injection, once a day for 7 days, once a month for 3 months)，Herombopag（10mg/d）+CsA(3-5 mg/kg/d, adjust the grain concentration 100-200ng/ml)
  Other Names: experimental
  Arms: rhTPO combined with Herombopag + CsA

SUMMARY:
Aplastic anemia (AA) is a group of clinical syndromes. Treatment options are very limited. The results of a previous clinical study showed good efficacy and a high safety profile of herombopag in improving thrombocytopenia, but this result needs to be supported by more data.

In our study, patients who were willing to participate in this study and were diagnosed with transfusion-dependent non-heavy aplastic anemia were randomized to the rhTPO combined with herombopag + cyclosporine group and given rhTPO (at a dose of 1500 U by subcutaneous injection once daily for 7 d, 28 d for 3 courses) +Herombopag(10 mg/day for 3 months) + cyclosporine (3-5 mg/kg/d for 3 months). -5 mg/kg/d for at least 6 months) and herombopag + cyclosporine (10 mg/day for 3 months) + cyclosporine (3-5 mg/kg/d for at least 6 months) in the herombopag+ cyclosporine group to observe the efficacy and safety.

DETAILED DESCRIPTION:
Aplastic anemia (AA) is a group of clinical syndromes caused by a significant decrease in bone marrow hematopoietic tissue from different etiologies, resulting in hematopoietic failure. The prevalence of AA in China is 7.4 per 1 million. It peaks in the 15-25 and 60+ age groups and is more common in men than women. Treatment options are very limited. The results of a previous clinical study showed good efficacy and a high safety profile of herombopag in improving thrombocytopenia, but this result needs to be supported by more data.

In our study, patients who were willing to participate in this study and were diagnosed with transfusion-dependent non-heavy aplastic anemia were randomized to the rhTPO combined with herombopag + cyclosporine group and given rhTPO (at a dose of 1500 U by subcutaneous injection once daily for 7 d, 28 d for 3 courses) +Herombopag(10 mg/day for 3 months) + cyclosporine (3-5 mg/kg/d for 3 months). -5 mg/kg/d for at least 6 months) and Herombopag + cyclosporine (10 mg/day for 3 months) + cyclosporine (3-5 mg/kg/d for at least 6 months) in the herombopag+ cyclosporine group to observe the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Clearly diagnosed untreated NSAA.
3. At least one of the following conditions was met at the time of enrollment: hemoglobin <90 g/L. Platelet <30×109/L, neutrophils <1.0×109/L.
4. Baseline liver and kidney function (ALT, AST, Cr) was less than 2 times the normal value.
5. No active infection; Not pregnant or breastfeeding.
6. Agree to sign the consent form.
7. The Eastern Cancer Collaboration Group (ECOG) score was 0-2.

Exclusion Criteria:

1. pancytopenia caused by other causes, such as myelodysplastic syndrome (MDS).
2. There is cytogenetic evidence of clonal hematologic bone marrow diseases (MDS, AML).
3. PNH clone ≥50%.
4. Had received hematopoietic stem cell transplantation (HSCT) before enrollment.
5. Immunosuppressive therapy such as ATG or cyclosporine use for more than 2 weeks.
6. Infection or bleeding that is not controlled by standard treatment.
7. Allergic to recombinant TPO or Hitrepopar.
8. Active HIV, HCV or HBV infection or cirrhosis or portal hypertension.
9. Any concomitant malignancy or local basal cell carcinoma of the skin within 5 years.
10. Previous history of thromboembolic events, heart attack or stroke (including antiphospholipid antibody syndrome) and current use of anticoagulants.
11. Women who are pregnant or nursing (lactation).
12. Have participated in other clinical trials within 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
ORR at 3 Months | Week 14
  After 3 months of treatment, ORR was calculated by measuring platelets, hemoglobin, neutrophils, and transfusion independence
ORR at 6 Months | Week 26
  After 6 months of treatment, ORR was calculated by measuring platelets, hemoglobin, neutrophils, and transfusion independence

SECONDARY OUTCOMES:
3 months of drug safety | Week 14
  Assessing the incidence and severity of adverse events; All adverse events that occur or worsen within 3 months of treatment will be reported
6 months of drug safety | Week 26
  Assessing the incidence and severity of adverse events; All adverse events that occur or worsen within 6 months of treatment will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: always
Access Criteria: email request